CLINICAL TRIAL: NCT01202630
Title: A Triple-blind, Randomized, Placebo-controlled, Multi-center Study on the Effect of BIO-K+ CL1285 for Prevention of Recurrent Clostridium Difficile Infection
Brief Title: BIO-K+ CL1285 for Prevention of Recurrent Clostridium Difficile Infection
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: The site is unable to recruit patients.
Sponsor: Bio-K Plus International Inc. (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 09-SUS-05-BIK-02
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Recurrent Clostridium Difficile Infection
Keywords: Clostridium difficile; diarrhea
MeSH Terms: conditions — Clostridium Infections; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental): BIO-K+ CL1285
  Interventions: Dietary Supplement: Lactobacillus acidophilus CL1285® and Lactobacillus casei
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus acidophilus CL1285® and Lactobacillus casei — 2 capsules of Lactobacillus acidophilus CL1285® and Lactobacillus casei (50 billion cfu/capsule), consumed once daily for 60 days
  Other Names: BIO-K+ CL 1285
  Arms: Probiotic
Dietary Supplement: Placebo — 2 capsules of placebo (no live cells), consumed once daily for 60 days
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of BIO-K+ CL1285 for prevention of recurrent Clostridium difficile infection.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Presence of two or more loose or liquid stools in the 24-hour period prior to initiation of antibiotic therapy
3. Hospitalized and starting antibiotic therapy for Clostridium difficile infection (CDI) or recurrent Clostridium difficile infection (RCDI), diagnosed with a positive stool culture
4. Agree to use contraception throughout study period, unless postmenopausal or surgically sterile (females only)
5. Understand the nature and purpose of the study including potential risks and side effects
6. Willing to comply with the requirements of the study

Exclusion Criteria:

1. History of 2 or more clostridium difficile infections at any time prior to the current episode
2. Presence of severe chronic and/or inflammatory condition
3. Impaired immunity, e.g. undergoing immunotherapy or chemotherapy
4. Major gastrointestinal complication, e.g. Crohn's disease or ulcer
5. Current treatment with nasogastric tube, ostomy, or parenteral nutrition
6. Use of proton pump inhibitors
7. Pregnant female or breastfeeding
8. Eating disorder
9. History of alcohol, drug, or medication abuse
10. Daily consumption of probiotics, fermented milk, and/or yogurt
11. Known allergies to any substance in the study product
12. Participation in another study with any investigational product within 3 months of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2010-06; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of recurrent Clostridium difficile infection | 60 days

SECONDARY OUTCOMES:
Duration of recurrent diarrhea episodes | 60 days
Presence of gastrointestinal symptoms | 60 days
Adverse events | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Cornelius J Foley, MD, Principal Investigator — Parker Jewish for Health Care and Rehabilitation
Locations (1):
- Parker Jewish Institute, New Hyde Park, New York, United States

REFERENCES:
- [Background] Gao XW, Mubasher M, Fang CY, Reifer C, Miller LE. Dose-response efficacy of a proprietary probiotic formula of Lactobacillus acidophilus CL1285 and Lactobacillus casei LBC80R for antibiotic-associated diarrhea and Clostridium difficile-associated diarrhea prophylaxis in adult patients. Am J Gastroenterol. 2010 Jul;105(7):1636-41. doi: 10.1038/ajg.2010.11. Epub 2010 Feb 9. PMID 20145608